CLINICAL TRIAL: NCT04982367
Title: A Prospective, Multicenter, Randomized Controlled Trial Comparing the Efficacy and Safety Between Sirolimus Coated Balloon Catheter and Paclitaxel Coated Balloon Catheter in the Treatment of Femoropopliteal Artery Stenosis.
Brief Title: Acoart SCB SFA: Sirolimus Coated Balloon Catheter in the Treatment of Femoropopliteal Artery Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acoart SCB SFA
Record Dates: First submitted 2021-07-21; First posted 2021-07-29 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Artery Disease
Keywords: Drug eluting balloon catheter; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus-eluting balloon angioplasty (Experimental): Using Sirolimus Coated Balloon Catheter in the treatment of stenosis or occlusion in superficial femoral artery(SFA) and/or popliteal artery
  Interventions: Device: Sirolimus-eluting balloon catheter
- Paclitaxel-eluting balloon angioplasty (Active Comparator): Using Paclitaxel Coated Balloon Catheter in the treatment of stenosis or occlusion in superficial femoral artery(SFA) and/or popliteal artery
  Interventions: Device: Paclitaxel-eluting balloon catheter

INTERVENTIONS:
Device: Sirolimus-eluting balloon catheter — Sirolimus-eluting balloon catheter designed and produced by Acotec
  Other Names: Sirolimus coated balloon catheter
  Arms: Sirolimus-eluting balloon angioplasty
Device: Paclitaxel-eluting balloon catheter — Paclitaxel-eluting balloon catheter (trade name:DHALIA)
  Other Names: Paclitaxel coated balloon catheter
  Arms: Paclitaxel-eluting balloon angioplasty

SUMMARY:
A prospective randomized trial designed to compare the efficacy and safety of Sirolimus coated balloon (SCB) versus paclitaxel coated balloon (DCB) in the treatment of femoropopliteal artery stenosis

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤80 years old
* Had lower extremity arterial occlusive diseases, and Rutherford classification is 2-5
* SFA and/or popliteal artery had severe stenosis (stenosis degree ≥70%) or occlusion.
* The length of target lesion less than 20 cm
* Subject (or legal guardian) understands the study requirements and procedures and provides written Informed Consent before any study tests or procedures are performed

Exclusion Criteria:

* The plasma creatinine level is higher than 150 umol/L
* Thrombolysis or thrombectomy is required
* There are more than 2 lesion need to treat in the target vessel.
* The patient had underwent lower-limb arterial surgery or thrombolysis on the target limb within 6 weeks.
* The target lesion had residual stenosis>30% or flow-limit dissection after pre-dilatation.
* The patient had outflow less than 1 vessel
* The lesion located in a stent.
* Patient has a known allergy to aspirin, clopidogrel, heparin, paclitaxel, sirolimus or contrast medium that cannot be adequately pre-medicated.
* Women who are pregnant or breast-feeding.
* The subjects have participated in other drug property studies or device studies that have not yet completed the main end point.
* Patient has life expectancy of less than 12 months.
* The investigator think the patient is not suitable for participation in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
The primary patency rate of target lesion at 12 months post-procedure | 12 months post-procedure
  Defined as freedom from clinically driven target lesion revascularization (CD-TLR) and binary restenosis (restenosis defined as duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥2.4)

SECONDARY OUTCOMES:
Rate of device success | immediate post-procedure
  Defined as successful delivery, balloon inflation, deflation and retrieval of the intact study device without burst below the rated burst pressure (RBP)
Rate of clinically driven target lesion revascularization (CD-TLR) at 12 months post-procedure | 12 months post-procedure
  Defined as any reintervention at the target lesion due to symptoms or the following index: drop of ABI >20% or ABI >0.15 compared to the post-procedure ABI during 12 months post-procedure
The change of Rutherford class from baseline | 12 months post-procedure
  Defined as change in target limb Rutherford class from baseline to 12 months
The change of ankle-brachial index (ABI) from baseline | 12 months post-procedure
  Defined as change of target limb ABI from baseline to 12 months
Rate of composite safety endpoint | 30 days post-procedure
  Defined a composite rate of device-related or procedure-related death, major target limb amputation (above-the-ankle amputation), clinically driven target lesion revascularization (CD-TLR) or target lesion thrombotic events through 30 days post- procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guo Wei, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China